CLINICAL TRIAL: NCT07332130
Title: Effect of Adding Dexmedetomidine to Bupivacain _fentanyl Mixture in Spinal Analgesia for Normal Labour
Brief Title: Spinal Analgesia in Labour Pain
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Minia University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Ragab Mohamed, residant, Minia University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1337/11/2024
Record Dates: First submitted 2025-12-02; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-10

CONDITIONS: Labour Analgesia

STUDY DESIGN:
Intervention Model Description: effect of adding dexmetomidine to bupivcain fentanyl mixture in spinal analgesia for normal labour
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Masking Description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DEX (Active Comparator): Participants receive intrathecaliy hyperbaric bupivacaine 2.5 mg (0.5 mL) combined with dexmedetomidine 2.5 µg and fentanyl 25 µg, diluted to a total volume of 2.5 mL. The solution will be administered as a single spinal injection under aseptic conditions.
  Interventions: Drug: injecting dexmedetomidine
- CONTROLLED (Active Comparator): Participants will receive intrathecaliy hyperbaric bupivacaine 2.5 mg (0.5 mL) combined with fentanyl 25 µg, diluted to a total volume of 2.5 mL. The solution will be administered as a single spinal injection under aseptic conditions.
  Interventions: Drug: injecting mixture of bupivacaine fentanyl

INTERVENTIONS:
Drug: injecting dexmedetomidine — injecting dexmedetomidine intrathecally during labour pain
  Arms: DEX
Drug: injecting mixture of bupivacaine fentanyl — injecting mixture of bupivacaine fentanyl intrathecally
  Arms: CONTROLLED

SUMMARY:
To evaluate the efficacy and safety of dexmedetomidine as an adjuvant to bupivacain and fentanyl in spinal Analgesia to decreases pain during normal labour

DETAILED DESCRIPTION:
Effect of adding dexmedetomidine to bupivacain fentanyl mixture in spinal analgesia for normal labour

ELIGIBILITY:
Inclusion Criteria:

Age of patint is between 18 and 40 years. gestational age of fetus is more than 37 weeks. singleton viable fetus and cephalic presentation. spontaneous labor with cervix dilation more than 5cm.

Exclusion Criteria:

Drug allergy. Blood Disease. Infection at site of injection. patient takes anticoagulants. patient has pre-eclampsia ,cardiac disease (NYHA III-IV) or diabetes mellitus type I prior to the pregnancy patients refuse

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-24 (Estimated); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
changes in numeric pain intensity score ( NPSI) maximum 10 minimum 0 | baseline
  evaluate the safety and effecacy of dexmetomidine for labour pain by numeric pain intensity score maximum 10 ( sever pain ), minimum 0 ( no pain )
duration of sensory blockade | 5 minutes after injection of analgesic agents till normal delivery done
  change in numeric pain intensity score ( NPIS )
changes in numeric pain intensity score ( NPIS ) | 5 minutes, 10 minutes, 15 minutes, 30 minutes and 45 minintes after injection of analgesic agents
  Scores range from 0-10 points, maximum ( 10 ) means sever pain, minimum ( 0 ) means no pain

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ragab, master, Principal Investigator — Minia University Hospitals
Locations (1):
- Minya, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD,
Supporting Information: Study Protocol
Time Frame: december 2025 - december 2026
Access Criteria: labour analgesia
URL: https://clinicaltrials.gov/